CLINICAL TRIAL: NCT03091439
Title: A Phase 2, Multicenter, Open-label, Randomized, Comparator-controlled Trial of the Safety and Efficacy of Dalbavancin Versus Active Comparator in Adult Patients With Osteomyelitis Known or Suspected to be Due to Gram-positive Organisms
Brief Title: Safety and Efficacy of Dalbavancin Versus Active Comparator in Adult Patients With Osteomyelitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision outlined by the corporation.
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3026-201-008
Record Dates: First submitted 2017-03-21; First posted 2017-03-27 (Actual); Results first posted 2018-09-26 (Actual); Last update posted 2018-09-26 (Actual); Status verified 2018-08

CONDITIONS: Osteomyelitis
Keywords: Osteomyelitis; dalbavancin; antibiotic
MeSH Terms: conditions — Osteomyelitis | interventions — dalbavancin; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dalbavancin (Experimental): Participants received Dalbavancin 1500 mg, intravenous (IV) administration over 30 minutes on Day 1 and on Day 8.
  Interventions: Drug: Dalbavancin
- Standard of Care (Active Comparator): Participants received an antibiotic consistent with standard of care (SOC) for osteomyelitis based on Investigator judgment. The duration of treatment will be 4-6 weeks.
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Dalbavancin — Participants received Dalbavancin 1500 mg, intravenous (IV) administration over 30 minutes on Day 1 and on Day 8.
  Other Names: Dalvance®; Xydalba™
  Arms: Dalbavancin
Drug: Standard of Care — Participants received an antibiotic consistent with standard of care (SOC) for osteomyelitis based on Investigator judgment. The duration of treatment was 4-6 weeks.
  Arms: Standard of Care

SUMMARY:
This clinical study will be a multi-center, randomized, open-label, active-controlled, parallel-group study comparing dalbavancin to standard of care (SOC) therapy in osteomyelitis.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of osteomyelitis (first episode) defined by:
* Pain or point tenderness upon palpation or probing to bone
* Plain radiograph or Magnetic resonance imaging (MRI) consistent with osteomyelitis (indistinctly marginated edema-like pattern of bone marrow hypointensity on unenhanced T1-weighted sequences, hyperintensity on fat-saturated T2-weighted and Short tau inversion recovery (STIR) sequences and/or abnormal enhancement on gadolinium-enhanced fat-saturated T2-weighted sequences, with or without visible periostitis or cortical bone destruction) OR Gram-positive cocci documented on a baseline Gram-stain from a bone specimen
* Elevated C-reactive protein (CRP) (low sensitivity) above the upper limit of normal (ULN) (reference range for low sensitivity CRP is 3-10 mg/L)
* Subjects must be willing and able, if discharged from the hospital, to return to the hospital or a designated clinic for scheduled visits, treatment, laboratory tests, and other outpatient procedures as required by the protocol.

Exclusion Criteria:

* Treatment with an investigational drug within 30 days preceding the first dose of investigational product.
* Receipt of > 24 hours of potentially effective IV antibacterial therapy for osteomyelitis within 96 hours of randomization, unless the pathogen isolated was documented to be Methicillin-resistant Staphylococcus aureus (MRSA) that was resistant to the administered antibiotic.
* A prior episode of osteomyelitis, or a failed course of therapy for osteomyelitis.
* Infection associated with a burn wound, with a sacral decubitus ulcer, or with multiple sites of osteomyelitis.
* Septic arthritis that is non-contiguous to osteomyelitis, as diagnosed by isolation of a pathogen from synovial fluid culture.
* Immunosuppression/immune deficiency
* Evidence of Gram-negative bacteria by Gram stain in the absence of Gram-positive organisms.
* Gram-negative bacteremia
* Patients with concomitant endocarditis, necrotizing fasciitis, or prosthetic material at the site of infection at the time of study initiation.
* Infection due to an organism known prior to study entry to not be susceptible to dalbavancin (dalbavancin mean inhibitory concentration [MIC] > 0.25 μg/mL) or vancomycin (vancomycin MIC > 2 μg/mL).
* Concomitant systemic antibacterial therapy for Gram-positive infections (eg, rifampin, gentamicin).
* Known or suspected hypersensitivity to glycopeptide antibiotics.
* Patients with a rapidly fatal illness, who are not expected to survive for 3 months.
* Pregnant or nursing females; positive urine (or serum) pregnancy test at Screening (pre-menopausal females only) or after admission (prior to dosing)
* Sexually active females of childbearing potential who are unwilling or unable to use an acceptable method of contraception from at least the first dose of study drug until the last pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Urania Rappo, MD, Study Director — Allergan
Locations (1):
- Midway Immunology and Research Center, Ft. Pierce, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Although this was a planned multi-center study, the study was terminated and only one investigative site in the United States enrolled a participant.
Period: Overall Study
Arm/Group | Dalbavancin | Standard of Care
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Study Terminated by the Sponsor | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Randomized Participants. 1 participant was enrolled in the Dalbavancin arm and 0 participants were enrolled in the Standard-of-Care arm. Due to confidentiality considerations, baseline data is not being provided to protect participant privacy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dalbavancin | Standard of Care | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical
Sex: Female, Male
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinical Response at Day 42 in the Clinically Evaluable (CE) Population
Description: Clinical response can be either cure, failure, or indeterminate. Cure was defined as recovery without need for additional antibiotic therapy. Failure was defined as the requirement of additional antibiotic therapy, new purulence, amputation due to progression of infection, requiring > 6 weeks of treatment in the SOC arm or death (for any reason). Indeterminate was defined as lost to follow-up or amputation due to vascular insufficiency. The number of participants in each response category is reported.
Time Frame: Day 42
Population: CE population included all participants in the mITT Population who received ≥ 1 dose of dalbavancin or ≥ 2 weeks of comparator and ≤ 1 dose of another (non-study) systemic antibiotic with activity against the causative organism for an indication other than osteomyelitis. No participants were enrolled in the SOC arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 1 | 0
Participants
  Cure | 1 | 0
  Failure | 0 | 0
  Indeterminate | 0 | 0

2. Secondary Outcome: Number of Participants With Clinical Improvement at Day 28 in the Modified Intent-to-Treat (mITT) Population
Description: Clinical improvement was based on an assessment of pain and/or point tenderness compared to Baseline and assessment of inflammation as measured by C-reactive Protein (CRP). Clinical improvement was defined as no worsening of pain from Baseline, if present, and improvement in inflammation.
Time Frame: Baseline (Day 0) to Day 28
Population: mITT population including all randomized participants who received randomized medication and met criteria for known or suspected Gram-positive osteomyelitis. Participants from whom only a Gram-negative pathogen was isolated from blood and/or bone culture were excluded. No participants were enrolled in the SOC arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 1 | 0
Participants | 1 |

3. Secondary Outcome: Number of Participants With Clinical Improvement at Day 28 in the CE Population
Description: as for outcome 2
Time Frame: Baseline (Day 0) to Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 1 | 0
Participants | 1 | 0

4. Secondary Outcome: Number of Participants With Clinical Response at Day 42 in the mITT Population
Description: Clinical response can be either cure, failure, or indeterminate. Cure was defined as recovery without need for additional antibiotic therapy. Failure was defined as the requirement of additional antibiotic therapy, new purulence, amputation due to progression of infection, requiring > 6 weeks of treatment in the SOC arm or death (for any reason). Indeterminate was defined as lost to follow-up or amputation due to vascular insufficiency.
Time Frame: Day 42
Population: mITT population included all randomized participants who received randomized medication and met the criteria for known or suspected Gram-positive osteomyelitis. Participants from whom only a Gram-negative pathogen was isolated from blood and/or bone culture were excluded. No participants were enrolled in the SOC arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 1 | 0
Participants
  Cure | 1 | 0
  Failure | 0 | 0
  Indeterminate | 0 | 0

5. Secondary Outcome: Number of Participants With Clinical Response at Day 42 in the Microbiological Modified Intent-to-Treat (Micro-mITT) Population
Description: as for outcome 4
Time Frame: Day 42
Population: micro-mITT included participants in the mITT Population with a Gram-positive pathogen isolated from blood and/or bone specimen. No participants met criteria for the micro-mITT population.
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Clinical Response at Day 180 in the mITT and CE Populations
Description: as for outcome 4
Time Frame: Day 180
Population: Due to early termination of the study prior to the Day 180 visit, the participant enrolled did not have data collected for this visit, but did have an early termination visit prior to Day 180.
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Number of Participants With Clinical Response at Day 365 in the mITT and CE Populations
Description: as for outcome 4
Time Frame: Day 365
Population: Due to early termination of the study prior to the Day 180 visit, the participant enrolled did not have data collected for the visits at Day 180 or Day 365, but did have an early termination visit prior to Day 180.
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants With Clinical Response by Pathogen at Day 42 in the CE Population
Description: as for outcome 4
Time Frame: Day 42
Population: There were no pathogens identified in this study; the participant enrolled had no pathogens detected on blood culture, and the optional bone biopsy was not performed.
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants With Clinical Response by Pathogen at Day 180 in the CE Population
Description: as for outcome 4
Time Frame: Day 180
Population: as for outcome 8
Arm/Group | Dalbavancin | Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline to last visit (Up to Day 108)
Description: No participants were enrolled in the SOC arm.
Arm/Group | Dalbavancin | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/39/NCT03091439/Prot_SAP_000.pdf